CLINICAL TRIAL: NCT05002699
Title: Investigating the Impact of Alzheimer's Disease Diagnostics in British Columbia (IMPACT-AD BC)
Brief Title: Investigating the Impact of Alzheimer's Disease Diagnostics in British Columbia
Acronym: IMPACT-AD BC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Brain Canada (Other); Health Canada (Other Government); Michael Smith Foundation for Health Research (Other); Women's Brain Health Initiative (Unknown); St. Paul's Foundation (Unknown)
Responsible Party: Principal Investigator, Mari L. DeMarco, PhD, Clinical Associate Professor, University of British Columbia
Other Study IDs: H17-01339
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease; Dementia; Cognitive Impairment; Mild Cognitive Impairment
Keywords: Biomarkers; Cerebrospinal fluid; Amyloid beta-Peptides; tau Proteins
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Alzheimer's disease CSF biomarkers — Measurement of amyloid beta peptide 1-42, amyloid beta peptide 1-40, and total tau in cerebrospinal fluid.

SUMMARY:
The 'Investigating the Impact of Alzheimer's Disease Diagnostics in British Columbia' (IMPACT-AD BC) study is an observational, longitudinal cohort study that will examine the impact of cerebrospinal fluid (CSF) testing for core Alzheimer's disease biomarkers on clinical decision making, diagnosis and health system utilization. In addition to data collection from physicians, the study will engage patients and their care partners in assessing the value of biomarker testing. IMPACT-AD BC investigators hypothesize that testing for CSF biomarkers of Alzheimer's disease in individuals with cognitive impairment, as part of routine clinical care, improves clinical management, diagnostic certainty, diagnostic accuracy, and healthcare resource utilization, and that patients and their care partners find the information valuable in planning for the future.

DETAILED DESCRIPTION:
The IMPACT-AD BC study is an observational, longitudinal cohort study designed to understand the impact of cerebrospinal fluid (CSF) testing for core Alzheimer's disease biomarkers on clinical decision making, diagnosis, health system utilization, and patients and their care partners.

Dementia specialists from multiple sites in the Canadian province of British Columbia will be approached to provide informed consent to participate. When these physicians order Alzheimer's disease CSF biomarker testing as part of routine care (DeMarco et al 2020), their patients will be eligible to participate in the study. Eligible patients (the patient participants) and their study partners (e.g., a family member or care partner) will be approached to provide informed consent to participate. The dementia specialists will provide diagnosis and management plans for their consenting patient participants before and after Alzheimer's disease CSF biomarker results. One year after release of the Alzheimer's disease CSF biomarker results, dementia specialists complete another questionnaire to assess the stability of their responses. In addition to these data, the study will collect patient participant/care partner perspectives on CSF biomarker testing post-results disclosure.

Via the IMPACT-AD BC study, the investigators will collect the first data of its kind on the utility of CSF biomarkers in routine care in Canada, with the overall goal of improving care and support systems for individuals living with neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participant is either a dementia specialist, or a patient of a consenting dementia specialist;
* Patient participant is age 40 and older;
* Patient participant has a diagnosis verified by a dementia specialist within 24 months of: subjective cognitive decline (Shaw et al., 2018), or mild cognitive impairment or dementia, according to DSM-IV (DSM-IV-TR, 2000) and/or National Institutes of Aging-Alzheimer's Association (Albert et al., 2011; McKhann et al., 2011) criteria;
* The etiologic cause of cognitive impairment is uncertain after a comprehensive evaluation by a dementia specialist, including general medical and neurological examination, mental status testing including standard measures of cognitive impairment, laboratory testing, and structural neuroimaging;
* Cognitive disorder is considered to be on the Alzheimer's continuum, including, but not limited to, mild cognitive impairment with suspected Alzheimer's pathology that does not reach the criteria for dementia;
* Dementia specialist deems that CSF Alzheimer's disease biomarkers are appropriate as per routine clinical care;
* Patient participant consents to a lumbar puncture for CSF analysis as part of clinical care.

Exclusion Criteria:

* Patient participant has normal cognition;
* Patient participant lumbar puncture requires imaging guidance;
* Knowledge of amyloid status, in the opinion of the treating dementia specialist, may cause significant psychological harm or otherwise negatively impact the patient or family;
* Amyloid status already known to patient or dementia specialist based on prior Aβ positron emission tomography (PET) imaging or previous CSF analysis;
* Aβ and tau CSF biomarkers ordered solely based on a family history of dementia, presence of apolipoprotein E4 genotype, or as a screening test for asymptomatic individuals;
* Aβ and tau CSF biomarkers ordered for non-medical purposes (e.g., legal, employment screening, insurance coverage, patient or family member curiosity);
* Current (i.e., active) patient participation in an anti-amyloid or anti-tau therapeutic trial;
* Presence of other significant chronic brain disease in patient (e.g., malignant tumor);
* Patient had symptomatic stroke or transient ischemic attack within the previous 12 months;
* Life expectancy of patient is less than 24 months based on medical co-morbidities;
* Lack of caregiver who can provide corroborative information if the patient participant lacks capacity to do so themselves.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient participants presenting with suspected preclinical, prodromal and Alzheimer's dementia, and meeting the appropriate use criteria for lumbar puncture and CSF biomarker testing (Shaw et al., 2018), will be enrolled along with their study partner and referring dementia specialist. A dementia specialist is defined as a self-identified physician trained and board-certified in neurology, psychiatry, or geriatric medicine who devotes a substantial proportion (≥ 25%) of patient contact time to the evaluation and care of adults with acquired cognitive impairment or dementia (Johnson et al., 2013).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of Alzheimer's disease core CSF biomarker testing on the management of patients meeting the appropriate use criteria for lumbar puncture and testing. | 12 months
  Determine the percent change between intended management (without biomarkers) and actual patient management (with biomarkers) in a composite measure of at least one of the following:
  1. Alzheimer's disease drug therapy;
  2. Other relevant drug therapy;
  3. Diagnostic procedure, imaging, other biofluid testing;
  4. Referral or counselling.
To describe the participant's experience with Alzheimer's disease CSF biomarker testing. | 6 months
  Describe the participant's experience with Alzheimer's disease CSF biomarker testing and evaluate the impact of testing on their planning and decision-making via interviews one-month and six-months post-disclosure of CSF biomarker results.
To describe the study partner's experience with Alzheimer's disease CSF biomarker testing. | 6 months
  Describe the study partner's experience with Alzheimer's disease CSF biomarker testing and evaluate the impact of testing on their planning and decision-making via interviews one-month and six-months post-disclosure of CSF biomarker results.

SECONDARY OUTCOMES:
To assess changes in participant management among various clinical presentations. | 12 months
  Describe the association of Alzheimer's disease CSF biomarker testing results with changes in management in individuals, from prodromal to dementia stage, presenting with typical clinical presentations of Alzheimer's disease versus atypical clinical presentations of Alzheimer's disease versus non-Alzheimer's neurodegenerative disorders.
To assess changes in participant management by clinical disease stage. | 12 months
  Describe the association of Alzheimer's disease CSF biomarker testing results with changes in management in individuals presenting with mild cognitive symptoms versus dementia.
To assess the impact of Alzheimer's disease core CSF biomarker testing on the change in diagnosis and diagnostic confidence. | 12 months
  Determine the percentage change in diagnosis and physician-rated diagnostic confidence from the pre-biomarker time-point to the post-biomarker time-point.

CONTACTS AND LOCATIONS:
Overall Officials: Mari L. DeMarco, PhD, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - Northern Health, Prince George, British Columbia
  - Providence Health Care, Vancouver, British Columbia
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Island Health, Victoria, British Columbia

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] DeMarco ML, Nguyen Q, Fok A, Hsiung GR, van der Gugten JG. An automated clinical mass spectrometric method for identification and quantification of variant and wild-type amyloid-beta 1-40 and 1-42 peptides in CSF. Alzheimers Dement (Amst). 2020 Jun 30;12(1):e12036. doi: 10.1002/dad2.12036. eCollection 2020. PMID 32617385
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders: DSM-IV [Internet]. 4th ed. Washington (DC): American Psychiatric Association; 1994 [cited 2010 Mar 8]. 866 p.
- [Background] Johnson KA, Minoshima S, Bohnen NI, Donohoe KJ, Foster NL, Herscovitch P, Karlawish JH, Rowe CC, Hedrick S, Pappas V, Carrillo MC, Hartley DM. Update on appropriate use criteria for amyloid PET imaging: dementia experts, mild cognitive impairment, and education. J Nucl Med. 2013 Jul;54(7):1011-3. doi: 10.2967/jnumed.113.127068. Epub 2013 Jun 10. PMID 23753186
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Shaw LM, Arias J, Blennow K, Galasko D, Molinuevo JL, Salloway S, Schindler S, Carrillo MC, Hendrix JA, Ross A, Illes J, Ramus C, Fifer S. Appropriate use criteria for lumbar puncture and cerebrospinal fluid testing in the diagnosis of Alzheimer's disease. Alzheimers Dement. 2018 Nov;14(11):1505-1521. doi: 10.1016/j.jalz.2018.07.220. Epub 2018 Oct 10. PMID 30316776
- See also: IMPACT-AD BC study website — https://www.impactAD.org/